CLINICAL TRIAL: NCT05732012
Title: Effectiveness of Online Sexual Health Psychoeducation Program Given to Physically Disabled Adolescents on Sexual Health Attitudes
Brief Title: The Effectiveness of the Sexual Health Psychoeducation Program for Physically Disabled Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Turkish Spinal Cord Paralysis Association (Unknown)
Responsible Party: Principal Investigator, Raife Aşık, Student, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sexual Health Psychoeducation
Record Dates: First submitted 2023-01-21; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Sexual Health; Adolescent; Physically Disabled; Psychological; Education
Keywords: Adolescent; Sexual health; Psychoeducation; Physically disabled; Sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Experimental): Interventions applied on Group-1 participants.
  Interventions: Behavioral: Sexual Health Psychoeducation Program
- Group-2 (No Intervention): No interventions applied on Group-2 participants.

INTERVENTIONS:
Behavioral: Sexual Health Psychoeducation Program — 62 adolescents were included in the study. Adolescents were assigned to intervention and control groups by randomization using simple numbers table. The intervention group was divided into 3 groups of 10 and included in a six-week psychoeducation program that lasted for one hour once a week, and 55 adolescents completed the program. The data on the sociodemographic characteristics of the adolescents constituting the sample were collected with the "Participant Information Form". Data on the effectiveness of the psychoeducation program on sexual health knowledge and attitudes were collected with the "Sexual Health Knowledge and Attitude Inventory" before the psychoeducation, at the end of the training and at the 3rd month of follow-up.
  Arms: Group-1

SUMMARY:
Objective: This research was planned to evaluate the effectiveness of the online psychoeducation program including sexual health education in physically disabled adolescents.

Materials and Methods: In this study, a randomized experimental design with pretest-posttest, follow-up measurement, intervention and control groups was used to evaluate the effectiveness of the sexual health online psychoeducation program in adolescents with physical disabilities. The universe of the study consists of adolescent members aged 12-15 in the Turkish Spinal Cord Paralysis Association.(N :600). Nearly 90 people with physical disabilities and their families, who were included in the inclusion criteria of the study, were reached through the institution. 62 people were included in the study as a result of the foresights made due to the intensity of their online classes due to the Covid- 19 pandemic, and their inability to volunteer for the subject of the research (they are ashamed and do not want to discuss it as a topic to be discussed). . Participants were divided into 31 participants as intervention group and 31 participants as control group by randomization method. The intervention group was divided into 3 groups of 10 and a six-week psychoeducation program lasting 60 minutes once a week was applied. At the end of the training, the intervention and control groups were given a post-test and a follow-up test at the end of the 3rd month.

DETAILED DESCRIPTION:
In addition to the nature of the adolescence period, which causes both physical and sexual differences and includes various difficulties, this period can be more complex for disabled adolescents. In addition to their physical problems, these adolescents try to make sense of their changing bodies and sexual identities, and according to studies, disabled adolescents may experience more psychosocial and psychosexual problems than adolescents without disabilities. Adolescents are expected to form sexual attitudes, values and engage in healthy sexual behaviors, as well as adapting to the functions of their changing and sexually maturing body. . Although sexual health education should have started within the family, families think that their adolescent children are not yet grown up and do not have a sexual life. In addition, it has been observed that the priority of families for their children is physical discomfort, and such developmental problems can be put in the background. This situation causes physically disabled adolescents to spend this process alone and cannot access sufficient information.

Psychoeducation applied in this study; meeting the sexual health education needs of the physically disabled; It is an online psychoeducation program designed to develop a positive attitude towards sexual health, increase adaptation to physical and emotional changes that may occur during adolescence, as well as the need for information. It is thought that the study can serve as a model for sexual health programs in adolescents with physical disabilities. This research was conducted to evaluate the effectiveness of the online psychoeducation program, which includes sexual health education, on sexual knowledge and attitudes in physically disabled adolescents.

The hypotheses of this study are:

H1. There is a significant difference between the post-test and follow-up total scores of the intervention group physically disabled adolescents compared to the pre-test total scores. It is expected that the control group scores will not differ.

H2. There is a significant difference between the post-test and follow-up test scores of the physically disabled adolescents in the intervention group and the post-test and follow-up test scores of the physically disabled adolescents in the control group in favor of the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 12-15
* Volunteering to participate in the research
* Not having a situation that prevents verbal communication
* Having and participating in online communication tools (computer, tablet, phone…)

Exclusion Criteria:

-Individuals with intellectual disabilities who have difficulty understanding and answering the research questions clearly and accurately. Not having online communication tools and not knowing how to participate (computer, tablet, phone…)

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Differentiation of Attitude Scores Regarding Sexually Transmitted Diseases by Groups | 4 month
Differentiation of Attitude Scores Regarding Sexuality According to Groups | 4 month
Differentiation of Attitude Scores Regarding Sexual Behaviors by Groups | 4 month
Differences in Attitude Scores Regarding Sexual Health and Personal Hygiene by Groups | 4 month
Differentiation of Attitude Scores Regarding Gender Roles by Group | 4 month
Differentiation of Attitude Scores Regarding Sexual Abuse by Groups | 4 month

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huurre T, Aro H.The psychosocial well-being of Finnish adolescents with visual impairments versus those with chronic conditions and those with no disabilities. Journal of Visual Impairment and Blindness.2000;94:625-637.
- [Background] Karaca S, Özaltın G. Experience with Structural Group Process: What Does a Group Process Executed with Blind Adolescents Teach?. Journal of Psychiatric Nursing. 2010; 1(2): 77-85.
- [Background] Greydanus DE, Pratt HD, Patel DR. Concepts of contraception for adolescent and young adult women with chronic illness and disability. Dis Mon. 2012 May;58(5):258-320. doi: 10.1016/j.disamonth.2012.02.001. PMID 22510362